CLINICAL TRIAL: NCT03796247
Title: Alexithymia Frequency and Interhemispheric Transfer in Patients With a First Demyelinating Event: Initial Phase of Multiple Sclerosis
Brief Title: Alexithymia Frequency and Interhemispheric Transfer in Patients With a First Demyelinating Event
Acronym: ALEXCIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2010_39; 2011-A00016-35 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Multiple Sclerosis
Keywords: cognition; alexithymia
MeSH Terms: conditions — Multiple Sclerosis; Affective Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- multiple sclerosis
- healthy control

SUMMARY:
Prevalence of alexithymia in multiple sclerosis (MS) is closed to 50% but is unknown in clinically isolated syndrome (CIS).The present study sought to characterize alexithymia in CIS patients and his link between psycho behavioral and cognitive disturbances.

In this context, the objectives of the present study were to (a ) define the prevalence of alexithymia in CIS patients, (b ) to study this relation between psycho behavioral and cognitive disorders frequently encountered in MS.

DETAILED DESCRIPTION:
The aim to recruit 40 CIS patients with at least two subclinical lesions on brain MRI. Patients are tested only one month at least after steroids intake and after 6 weeks at least after any relapse. The control group include 40 right -handed participants; each of them are matched for age, gender, and education level with a CIS patient.

The parameters to be evaluated are:

The prevalence of alexithymia is assessed by The Toronto Alexithymia Scale TAS-20, a self-reported scale. The TAS-20 total score corresponds to global level of alexithymia, as the sum of these three subdomains: 1.Difficulties in Identifying Feelings (DIF); 2. Difficulties in Describing Feelings (DDF); 3. Externally Oriented Thinking (EOT).

Standard neurological examination is performed by a neurologist using the Kurtzke Expanded Disability Status Scale (EDSS ).

The standardized neuropsychological battery, named BCcogSEP, is administrated. The BCcogSEP is made of eight tests commonly impaired in MS. Fourteen scores were obtained and a score was considered impaired when it was inferior to 5th percentile range compared to the normal range. The number of impaired scores are considered and a cognitive impairment is considered when 4 scores are superior or equal to percentile 5th.

For psychobehavioral assessments, the investigators estimated (a) depression (according to the Beck Depression Inventory; BDI (30)) and anxiety (according to the State-Trait Anxiety Inventory (31)); (b) apathy (according to the Lille Apathy Rating Scale (32)); (c) empathy (according to Interpersonal Reactivity Index; IRI).

ELIGIBILITY:
Inclusion Criteria:

* right-handed patient
* at least 1 month after steroid intake
* without severe neurological impairment
* without psychiatric disorder

Exclusion Criteria:

* patients with steroids in the last month
* patients with psychotropic drugs started in the last month
* patients with immunotherapies
* patients having contra indications for MRI
* pregnancy or breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: MS patients admited in MS center of Lille after the first neurological inflammatory clinical event
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2011-05-02 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency of alexithymia in the CIS population | Baseline: one session
  alexithymia is defined according to TAS-20 (Toronto Alexithymia Scale) The Toronto Alexithymia Scale is a measure of deficiency in understanding, processing, or describing emotions. The current version has twenty statements rated on a five-point Likert scale. ( range : Strongly disagree/Disagree/ Neither agree nor disagree/ Agree/ Strongly agree)

SECONDARY OUTCOMES:
relation between alexithymia and cognitive impairment in CIS patients and controls | Baseline: one session
  cognitive functions are evaluated by the standardized neuropsychological battery, named BCcogSEP. The BCcogSEP is made of eight tests commonly impaired in MS. Fourteen scores are obtained and a score is considered impaired when it is inferior to 5th percentile range compared to the normal range. The number of impaired scores is considered and a cognitive impairment is considered when 4 scores are superior or equal to percentile 5th.
relation between alexithymia and thymic disorder in CIS and controls | Baseline: one session
  Psychobehavioral assessments use the following Tools :
  We estimated depression according to the Beck Depression Inventory (BDI) The BDI consisted of twenty-one questions about how the subject has been feeling in the last week. Each question had a set of at least four possible responses, ranging in intensity. (0) I do not feel sad/ (1) I feel sad./ (2) I am sad all the time and I can't snap out of it/ (3) I am so sad or unhappy that I can't stand it.
  When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows:0-9: indicates minimal depression/ 10-18: indicates mild depression/ 19-29: indicates moderate depression/ 30-63: indicates severe depression.
relation between alexithymia and thymic disorder in CIS and controls | Baseline: one session
  Psychobehavioral assessments use the following Tools We estimated anxiety according to the State-Trait Anxiety Inventory (STAI) STAI is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis
relation between alexithymia and thymic disorder in CIS and controls | Baseline: one session
  Psychobehavioral assessments use the following Tools :
  We estimated apathy according to the Lille Apathy Rating Scale (LARS) The LARS is based on a structured interview. It includes 33 items, divided into nine domains. Responses are scored on a dichotomous scale
relation between alexithymia and thymic disorder in CIS and controls | Baseline: one session
  Psychobehavioral assessments use the following Tools :
  We estimated empathy according to Interpersonal Reactivity Index( IRI) The tool is a self-report comprising 28-items answered on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well".
to evaluate the callosal functions and inter-hemispheric transfer in CIS and controls | Baseline: one session
  dichotic listening tasks (number of sounds recognized from right or left ears) ; tactile localization recognition (number of right localization of right or left touch); letter matching test (number of right letter matching with right or left visual field) All those parameters are evaluated with qualitative assessment of functional MRI parameters

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Zephir, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France